CLINICAL TRIAL: NCT02868281
Title: The Effectiveness of Asthma Control Test Guided Treatment Compared With Usual Care in China Adult Asthma Patients
Brief Title: Asthma Control Test Guided Treatment in Chinese Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: MacroStat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201097
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Results first posted 2020-08-03 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Asthma
Keywords: Cluster Randomization; Peak Expiratory Flow; Forced Expiratory Volume; Standardized Asthma Quality of Life Questionnaire; Asthma Control Test
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects recruited at ACT centers (Experimental): For the subjects who will be recruited in the ACT centers, they will be treated based on the ACT score. If ACT score are = 25 for >=3 months then step-down the treatment; if ACT score >=20, <25 or ACT=25 for <3 months then there will be no change and if ACT score less than (<=) 19 then step-up the treatment.
  Interventions: Drug: ACT guided Routine Treatment
- Subjects recruited in the control centers (Active Comparator): For subjects who will be recruited in the control centers, they will be treated based on doctor's subjective judgment.
  Interventions: Drug: Routine Treatment

INTERVENTIONS:
Drug: ACT guided Routine Treatment — The ACT is a validated, short, easy to use, and self-administered instrument used to assess asthma control. Subjects in this group received routine treatment as per ACT score.
  Arms: Subjects recruited at ACT centers
Drug: Routine Treatment — Subjects in the controlled treatment group will receive usual care of asthma. This treatment was monitored and adjusted as usual by the patient's general practitioner.
  Arms: Subjects recruited in the control centers

SUMMARY:
This study is aimed to evaluate the effectiveness of Asthma Control Test (ACT) guided treatment compared with usual care in asthma subjects in China. It is designed to assist Chinese subjects and physicians improving adherence to the guidelines through the inclusion of the ACT in the patient's asthma management plan. This is a prospective, multicentre, cluster-randomized, open-label 24-week study. In this cluster-randomization design, each study center, considered as a cluster, will be randomized to either ACT guided treatment group or control group (usual care group). For the subjects who are recruited in the ACT centers, they will be treated based on the ACT score. If ACT score are equal to (=) 25 for more than equal to (>=) 3 months then the treatment will stepped-down; if ACT score >=20, less than (<) 25 or ACT=25 for <3 months then there will be no change and if ACT score less than (<=) 19 then the treatment will stepped-up. For subjects who are recruited in the control centers, they will be treated based on doctor's subjective judgment. Assignment to a treatment will not occur, as no treatment intervention is provided for this study. A total of 528 asthma subjects are planned in the study. The randomization will be stratified according to the Tier of the hospitals (Tier 3 verses Tier 2).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for study centre (clusters):

* General practice
* Located in Shanghai
* Providing asthma care

Inclusion Criteria for subject at Visit 0

* Age: 18 to 70 inclusive
* Gender: Male or Female
* Documented clinical history of asthma for at least 6 months prior to Visit 0
* At Visit 0, a demonstrable reversible increase in FEV1 of at least 12 percent (%) (and >=200 milliliter [mL]), 15 minutes after inhaling a short-acting bronchodilator or; at any time in the last 2 years documentary evidence of a reversible increase in FEV1 of at least 12% (and >=200 mL) 15 minutes after inhaling a short-acting bronchodilator; or demonstrable reversible increase in morning PEF of at least 15% (and >=200 mL) either spontaneously or after inhalation of a short-acting bronchodilator
* History of using inhaled corticosteroids alone or combined with an inhaled long-acting beta two agonist (LABA) treatment within 1 year prior to Visit 0
* Subjects must have an ACT score <20 at Visit 0
* Subject must have been able to read, comprehend, and record information in Chinese
* A signed and dated written informed consent must be obtained from the subject prior to study participation

Exclusion Criteria:

* History of Life-threatening asthma: Defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures within the last 6 months before Visit 0
* Subjects having severe and unstable asthma, with ACT score <12 at Visit 0, history of repeated severe exacerbations (3 per year) and/or a severe exacerbation in the previous 6 weeks before Visit 0.
* A current evidence of clinically significant uncontrolled medical condition or disease (e.g., psychological disorders, mental deficiency, severe hepatic and renal dysfunction, malignancy)
* Current smoker or ex-smoker with a more than 10 pack-year history of smoking
* Current clinically significant respiratory diseases other than asthma, (e.g., lung cancer, lung fibrosis, sarcoidosis, tuberculosis, chronic obstructive pulmonary disease)
* History of alcohol or medication abuse
* History of upper or lower respiratory tract infection within 4 weeks prior to Visit 0
* Enrolled in an asthma clinic or outpatient service in the past 12 months that provides comprehensive asthma management
* Subjects with a history of adverse reaction including immediate or delayed hypersensitivity to any intranasal, inhaled, or systemic corticosteroid and LABA therapy and to components of the inhalation powder (e.g., lactose) at Visit 0. In addition, subjects with a history of severe milk protein allergy that, in the opinion of the Investigator, contraindicates the subject's participation will also be excluded
* Females who are currently pregnant and lactating
* Subjects who have received any of the following medications in the 6 weeks preceding visit 0: oral/parenteral corticosteroids, oral beta two-agonists or slow-release bronchodilators, sodium cromoglycate or nedocromil sodium, ketotifen, anticholinergics, and anti-Immunoglobulin-E treatment
* Subjects who comply poorly with asthma treatment in the opinion of the investigator/inability or unwillingness to take asthma medication (non-compliance), follow directions or unable to complete a written paper daily record card and self-rating questionnaires
* Concurrently participating in another clinical study in which the subject is or will be exposed to an investigational or a non-investigational medication or device, or has participated in a clinical trial and has received an investigational product within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Subjects with contraindications to any asthma medications they will be taking during the study period, or whom should be excluded on account of the special warnings and precautions within the label of the asthma medication they are to be treated with during the study period
* Affiliation with Investigator Site: Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the afore mentioned that is involved in this study
* Subjects who plan to move away from the geographical area where the study is being conducted during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20843

REFERENCES:
- [Background] Ye L, Gao X, Tu C, Du C, Gu W, Hang J, Zhao L, Jie Z, Li H, Lu Y, Wang J, Jin X, Hu X, Wu S, Jin M. Comparative analysis of effectiveness of asthma control test-guided treatment versus usual care in patients with asthma from China. Respir Med. 2021 Jun;182:106382. doi: 10.1016/j.rmed.2021.106382. Epub 2021 Mar 30. PMID 33892217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 12 centers in China.
Pre-assignment Details: Total 583 participants were screened and 530 participants were enrolled into the study (53 participants were screen failures).
Groups:
- ACT Guided Treatment Group: Participants who were recruited in this Asthma Control Test (ACT) guided treatment group, were treated based on the ACT score. If ACT score =25 for >=3 months, then step-down treatment. If ACT score >=20 or <25 or ACT =25 for <3 months, then no change in treatment. If ACT score <=19, then step-up the treatment. ACT was completed prior to any other assessments were conducted.
- Usual Care Group: Participants who were recruited in this usual care group (control group), were treated based on physician's subjective judgement. Participants completed the ACT after investigator making the treatment decision, to ensure the investigator made treatment decision based on clinical judgement, not based on ACT score.
Period: Overall Study
Arm/Group | ACT Guided Treatment Group | Usual Care Group
Started | 252 | 278
Completed | 209 | 234
Not Completed | 43 | 44
Not completed — Adverse Event | 2 | 2
Not completed — Protocol Violation | 13 | 10
Not completed — Lost to Follow-up | 3 | 6
Not completed — Withdrawal by Subject | 11 | 15
Not completed — Physician Decision | 2 | 0
Not completed — Had protocol-defined asthma exacerbation | 8 | 8
Not completed — Inclusion/exclusion criteria violation | 3 | 2
Not completed — Long journey/moving away | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACT Guided Treatment Group | Usual Care Group | Total
Number analyzed (Participants) | 252 | 278 | 530
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.9 (12.74) | 48.1 (13.39) | 48.0 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 141 | 263
  Male | 130 | 137 | 267
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian-East Asian Heritage | 252 | 278 | 530

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had an ACT Total Score >=20 or an Improvement of More Than 3 Points in ACT During the 24-week Treatment Period
Description: ACT is a self-administered questionnaire comprising five items that were assessed on a five point categorical scale (1 to 5) and the scores are summed to give a total score ranging from 5 to 25, with a score of >=20 denoting 'well-controlled asthma', a score of 16-19 denoting 'not well-controlled asthma', and a score of <=15 denoting 'very poorly controlled asthma'. The total score was calculated as the sum of the scores from all 5 questions. Higher scores indicates improved asthma control. The recall period of the questionnaire was four weeks.
Time Frame: Up to Week 24
Population: Intent-To-Treat (ITT) Population consisted of all participants who signed informed consent form, were randomized and who had at least one post-Baseline assessment. Only those participants with data available at the specified data point were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | ACT Guided Treatment Group | Usual Care Group
Number analyzed (Participants) | 240 | 262
Percentage of participants | 99.2 | 94.3
Statistical Analysis 1: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.027, Mixed effect logistic regression; Odds Ratio (OR) = 7.87, 95% CI 2-sided [1.29 to 48.11] — The model included treatment, Baseline ACT total score, Baseline ACT total score squared, center, type of Baseline controller, gender and age, with the center as a random factor

2. Secondary Outcome: Mean Daytime Symptom Score Over the 24-week Treatment Period
Description: Participants recorded daytime asthma symptom scores in the daily record card (DRC). Any asthma-related symptoms, such as wheeze, shortness of breath, cough or chest tightness experienced during the previous 12 hours were rated as: 0= no symptoms during the day, 1= symptoms for one short period during the day, 2= symptoms for two or more short periods during the day, 3= symptoms for most of the day which did not affect daily activities, 4= symptoms for most of the day which did affect normal daily activities, 5= symptoms so severe that participant could not go to work or perform normal daily activities. Daytime symptom score was calculated by taking average of scores for all questions. The mean daytime asthma symptom score was calculated for each participant during the 4-weekly interval (Weeks 1-4, Weeks 5-8, Weeks 9-12, Weeks 13-16, Weeks 17-20 and Weeks 21-24) by taking average of 4 weeks. Score ranged from 0-5, higher scores indicates severe symptoms.
Time Frame: Weeks 1-4, Weeks 5-8, Weeks 9-12, Weeks 13-16, Weeks 17-20 and Weeks 21-24
Population: ITT Population. Only those participants with data available at the specified data point were analyzed (represented by n=x in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | ACT Guided Treatment Group | Usual Care Group
Number analyzed (Participants) | 236 | 259
Scores on a scale
  Weeks 1-4, n=236, 259 | 0.3 (0.05) | 0.4 (0.05)
  Weeks 5-8, n=227, 249: number analyzed (Participants) | 227 | 249
  Weeks 5-8, n=227, 249 | 0.2 (0.05) | 0.3 (0.05)
  Weeks 9-12, n=217, 240: number analyzed (Participants) | 217 | 240
  Weeks 9-12, n=217, 240 | 0.2 (0.05) | 0.2 (0.05)
  Weeks 13-16, n=210, 238: number analyzed (Participants) | 210 | 238
  Weeks 13-16, n=210, 238 | 0.1 (0.05) | 0.2 (0.05)
  Weeks 17-20, n=207, 233: number analyzed (Participants) | 207 | 233
  Weeks 17-20, n=207, 233 | 0.1 (0.05) | 0.2 (0.05)
  Weeks 21-24, n=205, 227: number analyzed (Participants) | 205 | 227
  Weeks 21-24, n=205, 227 | 0.1 (0.05) | 0.2 (0.05)
Statistical Analysis 1: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.222, Mixed Model Repeat Measures; Difference in Least Squares Mean = -0.1, 95% CI 2-sided [-0.2 to 0.0] — Weeks 1-4. The model included covariates of treatment, center, Baseline ACT total score, type of Baseline controller, gender, age and treatment-by-visit interaction, with the center as a random factor
Statistical Analysis 2: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.156, Mixed Model Repeat Measures; Difference in Least Squares Mean = -0.1, 95% CI 2-sided [-0.2 to 0.0] — Weeks 5-8. The model included covariates of treatment, center, Baseline ACT total score, type of Baseline controller, gender, age and treatment-by-visit interaction, with the center as a random factor
Statistical Analysis 3: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.245, Mixed Model Repeat Measures; Difference in Least Squares Mean = -0.1, 95% CI 2-sided [-0.2 to 0.0] — Weeks 9-12. The model included covariates of treatment, center, Baseline ACT total score, type of Baseline controller, gender, age and treatment-by-visit interaction, with the center as a random factor
Statistical Analysis 4: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.057, Mixed Model Repeat Measures; Difference in Least Squares Mean = -0.1, 95% CI 2-sided [-0.2 to 0.0] — Weeks 13-16. The model included covariates of treatment, center, Baseline ACT total score, type of Baseline controller, gender, age and treatment-by-visit interaction, with the center as a random factor
Statistical Analysis 5: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.151, Mixed Model Repeat Measures; Difference in Least Squares Mean = -0.1, 95% CI 2-sided [-0.2 to 0.0] — Weeks 17-20. The model included covariates of treatment, center, Baseline ACT total score, type of Baseline controller, gender, age and treatment-by-visit interaction, with the center as a random factor
Statistical Analysis 6: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.114, Mixed Model Repeat Measures; Difference in Least Squares Mean = -0.1, 95% CI 2-sided [-0.2 to 0.0] — Weeks 21-24. The model included covariates of treatment, center, Baseline ACT total score, type of Baseline controller, gender, age and treatment-by-visit interaction, with the center as a random factor

3. Secondary Outcome: Mean Night-time Symptom Score Over the 24-week Treatment Period
Description: Participants recorded night-time asthma symptom scores in the DRC. Any asthma-related symptoms, such as wheeze, shortness of breath, cough or chest tightness experienced during the previous 12 hours were rated as: 0= no symptoms during the night, 1= symptoms causing to wake once or wake early, 2= symptoms causing to wake twice or more (including waking early), 3= symptoms causing to be awake for most of the night, 4= symptoms so severe that participant did not sleep at all. Night-time symptom score was calculated by taking average of scores for all questions. The mean nighttime asthma symptom score was calculated for each participant during the 4 weekly interval (Weeks 1-4; Weeks 5-8, Weeks 9-12, Weeks 13-16, Weeks 17-20 and Weeks 21-24) by taking average of 4 weeks. Score ranged from 0-5, higher scores indicates severe symptoms.
Time Frame: Weeks 1-4, Weeks 5-8, Weeks 9-12, Weeks 13-16, Weeks 17-20 and Weeks 21-24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | ACT Guided Treatment Group | Usual Care Group
Number analyzed (Participants) | 236 | 258
Scores on a scale
  Weeks 1-4, n=236, 258 | 0.4 (0.07) | 0.5 (0.06)
  Weeks 5-8, n=226, 249: number analyzed (Participants) | 226 | 249
  Weeks 5-8, n=226, 249 | 0.3 (0.06) | 0.3 (0.06)
  Weeks 9-12, n=217, 240: number analyzed (Participants) | 217 | 240
  Weeks 9-12, n=217, 240 | 0.2 (0.06) | 0.3 (0.06)
  Weeks 13-16, n=209, 238: number analyzed (Participants) | 209 | 238
  Weeks 13-16, n=209, 238 | 0.2 (0.06) | 0.3 (0.06)
  Weeks 17-20, n=207, 233: number analyzed (Participants) | 207 | 233
  Weeks 17-20, n=207, 233 | 0.2 (0.06) | 0.2 (0.06)
  Weeks 21-24, n=205, 227: number analyzed (Participants) | 205 | 227
  Weeks 21-24, n=205, 227 | 0.2 (0.06) | 0.2 (0.06)
Statistical Analysis 1: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.487, Mixed Model Repeat Measures; Difference in Least Squares Mean = -0.05, 95% CI 2-sided [-0.18 to 0.09] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.546, Mixed Model Repeat Measures; Difference in Least Squares Mean = -0.04, 95% CI 2-sided [-0.16 to 0.09] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.314, Mixed Model Repeat Measures; Difference in Least Squares Mean = -0.06, 95% CI 2-sided [-0.17 to 0.06] — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.197, Mixed Model Repeat Measures; Difference in Least Squares Mean = -0.07, 95% CI 2-sided [-0.19 to 0.04] — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.282, Mixed Model Repeat Measures; Difference in Least Squares Mean = -0.06, 95% CI 2-sided [-0.17 to 0.06] — [estimate comment as in outcome 2, analysis 5]
Statistical Analysis 6: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.543, Mixed Model Repeat Measures; Difference in Least Squares Mean = -0.03, 95% CI 2-sided [-0.15 to 0.08] — [estimate comment as in outcome 2, analysis 6]

4. Secondary Outcome: Mean Change From Baseline in Forced Expiratory Volume in One Second (FEV1) at Week 24
Description: FEV1 is defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 was measured by spirometry. Baseline was defined as value at Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and at Week 24
Population: ITT Population. Only those participants with data available at the specified data point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | ACT Guided Treatment Group | Usual Care Group
Number analyzed (Participants) | 208 | 227
Liters | 0.159 (0.0573) | 0.098 (0.0559)
Statistical Analysis 1: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.273, Mixed Model Repeat Measures; Difference in Least Squares Mean = 0.060, 95% CI 2-sided [-0.059 to 0.180] — The model included covariates of treatment, center, Baseline FEV1, type of Baseline controller, gender and age, with the center as a random factor

5. Secondary Outcome: Mean Morning (Ante Meridiem [AM]) Peak Expiratory Flow (PEF) Over the 24-week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. Participants were provided with a Mini-Wright Peak Flow Meter and were taught how to measure and record their PEF. Participants recorded on DRC the best of three PEF measurements, using a Mini-Wright peak flow meter in the morning (7:00 to 10:00 AM) before taking any asthma drug. Mean AM PEF was calculated for each participant during the 4-weekly interval (Weeks 1-4; Weeks 5-8, Weeks 9-12, Weeks 13-16, Weeks 17-20 and Weeks 21-24) by taking average of 4 weeks.
Time Frame: Weeks 1-4, Weeks 5-8, Weeks 9-12, Weeks 13-16, Weeks 17-20 and Weeks 21-24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | ACT Guided Treatment Group | Usual Care Group
Number analyzed (Participants) | 239 | 261
Liters per minute
  Weeks 1-4, n=239, 261 | 340.4 (13.37) | 352.4 (13.03)
  Weeks 5-8, n=228, 251: number analyzed (Participants) | 228 | 251
  Weeks 5-8, n=228, 251 | 355.5 (13.39) | 362.7 (13.05)
  Weeks 9-12, n=220, 241: number analyzed (Participants) | 220 | 241
  Weeks 9-12, n=220, 241 | 362.2 (13.42) | 366.9 (13.08)
  Weeks 13-16, n=211, 239: number analyzed (Participants) | 211 | 239
  Weeks 13-16, n=211, 239 | 364.6 (13.40) | 367.9 (13.06)
  Weeks 17-20, n=207, 235: number analyzed (Participants) | 207 | 235
  Weeks 17-20, n=207, 235 | 366.0 (13.38) | 371.0 (13.04)
  Weeks 21-24, n=206, 229: number analyzed (Participants) | 206 | 229
  Weeks 21-24, n=206, 229 | 367.0 (13.43) | 371.0 (13.08)
Statistical Analysis 1: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.367, Mixed Model Repeat Measures; Difference in Least Squares Mean = -12.0, 95% CI 2-sided [-40.3 to 16.3] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.587, Mixed Model Repeat Measures; Difference in Least Squares Mean = -7.2, 95% CI 2-sided [-35.5 to 21.2] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.721, Mixed Model Repeat Measures; Difference in Least Squares Mean = -4.7, 95% CI 2-sided [-33.1 to 23.7] — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.801, Mixed Model Repeat Measures; Difference in Least Squares Mean = -3.3, 95% CI 2-sided [-31.7 to 25.1] — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.704, Mixed Model Repeat Measures; Difference in Least Squares Mean = -5.0, 95% CI 2-sided [-33.3 to 23.4] — [estimate comment as in outcome 2, analysis 5]
Statistical Analysis 6: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.762, Mixed Model Repeat Measures; Difference in Least Squares Mean = -4.0, 95% CI 2-sided [-32.4 to 24.5] — [estimate comment as in outcome 2, analysis 6]

6. Secondary Outcome: Mean Evening (Post Meridiem [PM]) PEF Over the 24-week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. Participants were provided with a Mini-Wright Peak Flow Meter and were taught how to measure and record their PEF. Participants recorded on DRC the best of three PEF measurements, using a Mini-Wright peak flow meter in the evening (6:00 to 9:00 PM) before taking any asthma drug. Mean PM PEF was calculated for each participant during the 4-weekly interval (Weeks 1-4; Weeks 5-8, Weeks 9-12, Weeks 13-16, Weeks 17-20 and Weeks 21-24) by taking average of 4 weeks.
Time Frame: Weeks 1-4, Weeks 5-8, Weeks 9-12, Weeks 13-16, Weeks 17-20 and Weeks 21-24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | ACT Guided Treatment Group | Usual Care Group
Number analyzed (Participants) | 239 | 261
Liters per minute
  Weeks 1-4, n=239, 261 | 342.2 (13.55) | 354.9 (13.22)
  Weeks 5-8, n=228, 251: number analyzed (Participants) | 228 | 251
  Weeks 5-8, n=228, 251 | 356.2 (13.60) | 364.6 (13.27)
  Weeks 9-12, n=220, 241: number analyzed (Participants) | 220 | 241
  Weeks 9-12, n=220, 241 | 362.7 (13.63) | 367.7 (13.29)
  Weeks 13-16, n=211, 239: number analyzed (Participants) | 211 | 239
  Weeks 13-16, n=211, 239 | 365.8 (13.61) | 368.9 (13.27)
  Weeks 17-20, n=207, 235: number analyzed (Participants) | 207 | 235
  Weeks 17-20, n=207, 235 | 366.9 (13.60) | 370.9 (13.26)
  Weeks 21-24, n=206, 229: number analyzed (Participants) | 206 | 229
  Weeks 21-24, n=206, 229 | 368.1 (13.67) | 372.0 (13.33)
Statistical Analysis 1: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.354, Mixed Model Repeat Measures; Difference in Least Squares Mean = -12.8, 95% CI 2-sided [-42.1 to 16.5] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.538, Mixed Model Repeat Measures; Difference in Least Squares Mean = -8.4, 95% CI 2-sided [-37.8 to 21.0] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.716, Mixed Model Repeat Measures; Difference in Least Squares Mean = -5.0, 95% CI 2-sided [-34.4 to 24.5] — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.822, Mixed Model Repeat Measures; Difference in Least Squares Mean = -3.1, 95% CI 2-sided [-32.5 to 26.3] — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.767, Mixed Model Repeat Measures; Difference in Least Squares Mean = -4.0, 95% CI 2-sided [-33.4 to 25.4] — [estimate comment as in outcome 2, analysis 5]
Statistical Analysis 6: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.779, Mixed Model Repeat Measures; Difference in Least Squares Mean = -3.8, 95% CI 2-sided [-33.4 to 25.7] — [estimate comment as in outcome 2, analysis 6]

7. Secondary Outcome: Mean Change From Baseline in Standardized Asthma Quality of Life Questionnaire (AQLQ[S]) Total Score at Week 24
Description: The AQLQ(S) contains 32 items in four domains: activity limitation (11 items), symptoms (12 items), emotional function (5 items) and environmental stimuli (4 items). Participant's response to each question was rated on a seven-point scale (1 to 7) where a value of 1 indicates "total impairment" and a value of 7 indicates "no impairment". The total AQLQ(S) score is calculated as the mean of all 32 items in the questionnaire. Hence, the total AQLQ(S) score ranged from 1 to 7 with higher scores indicating a higher quality of life. A change in score of greater than 0.5 can be considered clinically important. Baseline was defined as value at Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and at Week 24
Population: ITT Population. Only those participants with data available at the specified data point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | ACT Guided Treatment Group | Usual Care Group
Number analyzed (Participants) | 202 | 231
Scores on a scale | 1.5 (0.13) | 1.2 (0.13)
Statistical Analysis 1: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.059, Mixed Model Repeat Measures; Difference in Least Squares Mean = 0.3, 95% CI 2-sided [-0.0 to 0.6] — The model included covariates of treatment, center, Baseline AQLQ(S) score, type of Baseline controller, gender and age, with the center as a random factor

8. Secondary Outcome: Time to First ACT Score >=20 or Improvement of More Than 3 Points in ACT Over the 24-week Treatment Period
Description: ACT is a self-administered questionnaire comprising five items that were assessed on a five point categorical scale (1 to 5) and the scores are summed to give a total score ranging from 5 to 25, with a score of >=20 denoting 'well-controlled asthma', a score of 16-19 denoting 'not well-controlled asthma', and a score of <=15 denoting 'very poorly controlled asthma'. Higher scores indicates improved asthma control. The recall period of the questionnaire was four weeks. Median and inter-quartile range (first and third quartiles) are presented for time to first ACT score >=20 or improvement of more than 3 points in ACT over the 24-week treatment period.
Time Frame: Up to Week 24
Population: ITT Population. Only those participants with data available at the specified data point were analyzed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | ACT Guided Treatment Group | Usual Care Group
Number analyzed (Participants) | 229 | 224
Days | 33.0 [29.0 to 57.0] | 55.0 [29.0 to 98.0]
Statistical Analysis 1: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.010, Cox proportional hazards model; Hazard Ratio (HR) = 1.843, 95% CI 2-sided [1.160 to 2.926] — The model included treatment, Baseline ACT total score, center, type of Baseline controller, gender and age as covariates

9. Other Pre Specified Outcome: Annualized Rate of Moderate to Severe Asthma Exacerbation During 24-week Treatment Period
Description: Exacerbations were assessed by the physician at each scheduled visit by reviewing the DRC, as well as specific questioning on adverse events. A moderate asthma exacerbation was defined as a deterioration in asthma requiring treatment with an oral corticosteroid. Individual courses of oral corticosteroids were classified as separate exacerbations only if they were administered more than 1 week apart. Any course started within one week of finishing the previous course was considered part of the previous exacerbation. A severe asthma exacerbation was defined as a deterioration in asthma which requires hospital admission. Annualized Rate of moderate to severe asthma exacerbation during 24-week treatment period is presented.
Time Frame: Up to Week 24
Population: ITT Population. Only those participants with data available at the specified data point were analyzed.
Measure: Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | ACT Guided Treatment Group | Usual Care Group
Number analyzed (Participants) | 241 | 263
Exacerbations per year | 0.10 [0.04 to 0.25] | 0.09 [0.04 to 0.22]
Statistical Analysis 1: Comparison: ACT Guided Treatment Group vs Usual Care Group; Test type: Other; p = 0.897, Generalised linear model; Rate Ratio = 1.09, 95% CI 2-sided [0.32 to 3.73] — The model included treatment, Baseline ACT total score, type of Baseline controller, gender and age as covariates

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (AEs) and serious AEs were collected from start of study treatment (Day 1) up to Week 24
Description: Non-serious AEs and serious AEs were collected for Safety Population which consisted of all participants who were enrolled into the study and who had at least one DRC assessment.
Arm/Group | ACT Guided Treatment Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 1/252 | 0/278
Serious Adverse Events (participants affected / at risk) | 9/252 | 14/278
Other Adverse Events (participants affected / at risk) | 82/252 | 123/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACT Guided Treatment Group (N=252) | Usual Care Group (N=278)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0
Otitis media chronic (Infections and infestations) | 1 | 0
Salpingitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pelvic adhesions (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hypertrophic anal papilla (Gastrointestinal disorders) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0
Subclavian artery occlusion (Vascular disorders) | 0 | 1
Branchial cleft sinus (Congenital, familial and genetic disorders) | 0 | 1
Macular oedema (Eye disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACT Guided Treatment Group (N=252) | Usual Care Group (N=278)
Upper respiratory tract infection (Infections and infestations) | 18 | 47
Rhinitis (Infections and infestations) | 6 | 3
Nasopharyngitis (Infections and infestations) | 4 | 4
Bronchitis (Infections and infestations) | 3 | 16
Conjunctivitis (Infections and infestations) | 3 | 3
Respiratory tract infection (Infections and infestations) | 3 | 6
Urinary tract infection (Infections and infestations) | 3 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Otitis media (Infections and infestations) | 2 | 1
Pelvic inflammatory disease (Infections and infestations) | 2 | 0
Vaginal infection (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 1
Pulpitis dental (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tinea cruris (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Urethritis (Infections and infestations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Dysbacteriosis (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Gingival swelling (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Breath odour (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 4
Chest discomfort (General disorders) | 4 | 1
Chest pain (General disorders) | 2 | 2
Discomfort (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 4
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Tooth injury (Injury, poisoning and procedural complications) | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Endometrial thickening (Reproductive system and breast disorders) | 1 | 0
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0
Pelvic fluid collection (Reproductive system and breast disorders) | 1 | 0
Breast hyperplasia (Reproductive system and breast disorders) | 0 | 2
Palpitations (Cardiac disorders) | 1 | 2
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Adrenal mass (Endocrine disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0
Scleritis (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Vitreous opacities (Eye disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myofascitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 2 | 4
Dizziness (Nervous system disorders) | 1 | 2
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 1
Poor quality sleep (Nervous system disorders) | 0 | 1
Vascular headache (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urate nephropathy (Renal and urinary disorders) | 1 | 0
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 2
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 3
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-06-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT02868281/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT02868281/SAP_001.pdf